CLINICAL TRIAL: NCT06923189
Title: Efficacy Testing of a Multi-Level Family Planning Intervention to Increase Contraceptive Use and Reduce Unintended Pregnancy in Low Resource Settings
Brief Title: Efficacy Testing of a Multi-Level Family Planning Intervention
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); San Diego State University (Other); Yale University (Other); University of North Carolina, Chapel Hill (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 25.018.01; R01HD113806 (NIH)
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Unintended Pregnancy; Family Planning
Keywords: Unintended pregnancy; Contraceptive use; Family planning; Intervention; Cluster randomized controlled trial; Uganda; Couples
MeSH Terms: interventions — Water; Sanitation; Hygiene; Therapeutic Irrigation; Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Data collectors (interviewers)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Family Health = Family Wealth (Experimental): This arm receives the Family Health = Family Wealth intervention.
  Interventions: Behavioral: Family Planning Intervention
- Time- and attention-matched WASH intervention (Active Comparator): This arm receives an attention-matched comparator intervention focused on water, sanitation, and hygiene (WASH).
  Interventions: Behavioral: Water, Sanitation, and Hygiene (WASH) Intervention

INTERVENTIONS:
Behavioral: Family Planning Intervention — This multilevel intervention is comprised of community dialogues, or facilitated discussions, aimed to reshape community norms around gender roles, equity, and family size, and critically analyze the social and community influences of "family-wealth" and poverty with the overall goal of reconstructing individual attitudes and group norms on paths to/definitions of a "successful family" inclusive of family planning. Dialogues are enhanced to address knowledge, motivation, self-efficacy, and relationship dynamics, tailored to men and women. Sessions include both gender segregated and integrated groups with couples in the community. The intervention is paired with health system strengthening elements implemented with the intervention health clinics (provider training, strengthening skip the queue policies, linkage of family planning services directly to dialogues).
  Arms: Family Health = Family Wealth
Behavioral: Water, Sanitation, and Hygiene (WASH) Intervention — This intervention serves as the attention-matched control. The format and delivery will mirror that of the "Family Health = Family Wealth" intervention (i.e., number, timing, and duration of sessions). The focus of the intervention is on community sanitation and at-home hygiene (handwashing, food preparation) following an intervention manual that was developed for community groups in East Africa and tailored to the local Uganda context.
  Arms: Time- and attention-matched WASH intervention

SUMMARY:
The goal of this cluster randomized controlled trial is to learn if the multi-level, community-based family planning intervention, known as the Family Health=Family Wealth (FH=FW) program, can improve family planning outcomes in couples of reproductive age in Uganda. The main questions it aims to answer are:

1. Does FH=FW participation reduce unintended pregnancy and increase contraceptive uptake among couples who say they want to delay pregnancy over 24-months?
2. Does FH=FW participation reduce discontinuation of contraceptive methods for those who adopt them over 24-months?
3. What factors affect the implementation of the FH=FW intervention?

Researchers will compare change in the above outcomes in couples receiving the FH=FW intervention to those who instead receive a water, sanitation, and hygiene intervention.

Couples in the FH=FW arm will be asked to attend 6 groups sessions where they learn about family planning's benefits to their health and well-being alongside content to increase their shared spousal decision-making and communication skills, their access to family planning services, and their perceptions of community acceptance of family planning.

DETAILED DESCRIPTION:
In 2022, 29.7% of married women of reproductive age had an unmet need for family planning in Uganda, meaning they wanted to avoid pregnancy but were not using a modern contraceptive method. Filling the unmet need for family planning has important public health implications, including reductions in pregnancy-related health risks and deaths, and infant mortality. On the supply-side, community platforms to deliver family planning, as well as provider capacity to provide effective methods, need to be strengthened, but such efforts will not be optimized without addressing multilevel demand-side barriers to contraceptive use. Misinformation and fear of contraceptive side-effects, relationship dynamics, peer and family influence, and broader community norms promoting large family size and traditional gender roles influence family planning. This study will test the Family Health=Family Wealth (FH=FW) multi-level, community-based intervention, which employs health system strengthening efforts alongside transformative community dialogues to alter individual attitudes and the perception of community norms that discourage family planning. Community dialogues are delivered to groups of couples over 6-sessions enhanced to simultaneously address individual and interpersonal-level determinants of family planning and serve as a platform for community-based family planning and linkage to facility-based family planning services. The study aims are to: (1) In a cluster randomized trial, compare the efficacy of the FH=FW intervention vs. a time/attention matched comparator intervention at increasing modern contraceptive use and reducing unintended pregnancy among couples with an unmet need for family planning through 24-months, and identify potential mediators of the intervention effect. (2) Determine the intervention's effect on, and determinants of, contraceptive continuation. (3) Through a mixed-methods process evaluation, explore factors affecting the implementation of the intervention in order to improve feasibility, acceptability, and the likelihood of future adoption and sustainment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 (or emancipated minors - those 15-17 who are married and/or have children) to 49 and men aged 18 (or emancipated minors age 15-17) to 54. The upper age limits follow those used by the Demographic and Health Surveys (DHS) to define "reproductive age."
* Married or considers themselves married and living together most of the time
* Residing in communities selected for study inclusion
* Luganda speaking
* Sexually active with spouse within the past 3 months or planning to resume sex within the next 3 months if the woman is within 2 months postpartum
* Not currently pregnant (confirmed via pregnancy test); can be eligible to enroll later once postpartum
* The woman has an unmet need for family planning, i.e., the woman reports not wanting to become pregnant within the next 2 years but is not using any effective methods (IUD, injection, oral pill, implant, vasectomy, tubal ligation, condoms 90% of the time or more) or is using only lower-efficacy methods (condoms less than 90% of the time, lactational amenorrhea, fertility-awareness based methods e.g., counting method, withdrawal).

Exclusion Criteria:

* At least one person in the couple does not expect to be available for all sessions
* The woman or man is not able to reproduce due to a known medical reason (e.g., hysterectomy, as told by a doctor) or last period greater than 6 months for women that are not postpartum.

Ages: 15 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1464 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in modern contraceptive use among those with an unmet need for family planning | 4-, 8-, 12-, 16-, 20-, 24-months
  Proportion of couples where the woman currently wants to prevent pregnancy reporting modern contraceptive use.
  Measured through structured timeline follow-back (TLFB) interviews, which use cued recall techniques, e.g., identifying key dates to serve as anchors, to assess contraceptive use by week for the prior four-month period (used y/n, method). Pregnancy intentions (desire to prevent pregnancy) are reassessed and accounted for at each follow-up.
Unintended pregnancy incidence | 8-, 16-, 24-months
  Unintended pregnancy incidence (Yes/No) over 24 months. Measured through urine Human Chorionic Gonadotropin rapid pregnancy tests; classified as unintended if reporting they wanted to wait until later or not get pregnant at all at the time of the pregnancy test, captured through a Demographic and Health Survey item.

SECONDARY OUTCOMES:
Change from baseline in modern contraceptive use | 4-, 8-, 12-, 16-, 20-, 24-months
  Proportion of couples reporting modern contraceptive use in the full sample, regardless of pregnancy intentions.
  Measured through structured timeline follow-back (TLFB) interviews, which use cued recall techniques, e.g., identifying key dates to serve as anchors, to assess contraceptive use by week for the prior four-month period (used y/n, method).
Change from baseline in contraceptive autonomy | 4-, 8-, 12-, 16-, 20-, 24-months
  Proportion of women reporting contraceptive autonomy (y/n). Contraceptive autonomy (yes) is defined as those that want to delay pregnancy with modern contraceptives reporting contraceptive use or that do not want to delay pregnancy with modern contraceptives that are not using a method (positive outcome).
  Contraceptive autonomy (no) is defined as those not using a modern method when wanting to delay pregnancy with a modern method or using a method when not wanting to delay pregnancy are considered not having contraceptive autonomy.
  Contraceptive use is measured through structured timeline follow-back (TLFB) interviews, which use cued recall techniques, e.g., identifying key dates to serve as anchors, to assess contraceptive use by week for the prior four-month period (used y/n, method).
Change from baseline in contraceptive continuation rate | 4-, 8-, 12-, 16-, 20-, 24-months
  Duration of continuation: The time from starting contraceptive use to discontinuation (a period of discontinuation of 1 month or more).
  Contraceptive use is measured through structured timeline follow-back (TLFB) interviews, which use cued recall techniques, e.g., identifying key dates to serve as anchors, to assess contraceptive use by week for the prior four-month period (used y/n, method).

OTHER OUTCOMES:
Change from baseline in any contraceptive use among those with an unmet need for family planning | 4-, 8-, 12-, 16-, 20-, 24-months
  Proportion of couples where the woman currently wants to prevent pregnancy reporting any contraceptive use (included natural methods). Measured through structured timeline follow-back (TLFB) interviews, which use cued recall techniques, e.g., identifying key dates to serve as anchors, to assess contraceptive use by week for the prior four-month period (used y/n, method). Pregnancy intentions (desire to prevent pregnancy) are reassessed and accounted for at each follow-up.
Change from baseline in knowledge of contraceptives | 8-, 16-, 24-months
  Scale from the Uganda Demographic and Health Survey (DHS) aimed to assess knowledge of modern contraceptive methods; collected through interviewer-administered questionnaire. Possible range 0-1, greater scores indicate more knowledge.
Change from baseline in family planning attitudes | 8-, 16-, 24-months
  Family planning attitudes scale developed for use in Uganda to assess how participants would feel about using contraceptive methods; collected through interviewer-administered questionnaire. Scores range from 0-4 with greater scores indicating more positive attitudes towards family planning.
Change from baseline in perceived family planning norms | 8-, 16-, 24-months
  Scale adapted from the Family Planning Approval Index to assess the perceived acceptance of family planning and contraceptive use among partner, family, peers, and broader community; collected through interviewer-administered questionnaire. Scores range from 0-1 with greater scores indicating more positive perceived attitudes towards family planning among others.
Change from baseline in family planning intentions | 8-, 16-, 24-months
  Family planning intentions scale developed for use in Uganda to assess participants' plans to use contraceptives and family planning services in the future; collected through interviewer-administered questionnaire. Scores range between 0-4 with higher scores indicating greater intentions to use family planning services in the future.
Change from baseline in desired number of children (fertility desires) | 8-, 16-, 24-months
  Item from the Uganda Demographic and Health Survey (DHS) on the participants' fertility desires (i.e., desired number of additional children); collected through interviewer-administered questionnaire. This is a count variable that could range from zero upward (no limit).
Change from baseline in joint household decision-making | 8-, 16-, 24-months
  Joint household decision-making was measured with items from the Uganda DHS that ask respondents who primarily decides on: 1) how the money they earn is used; 2) how their spouses' earnings are used; 3) decisions about healthcare for yourself; and 4) decisions about major household purchases. Response options coded as self and partner jointly (1) vs. all other (0). Greater scores indicating more joint decision-making (range 0-1).
Change from baseline in gender inequitable attitudes | 8-, 16-, 24-months
  The mean of the 24-item Gender Equitable Men scale measured endorsement of traditional gender norms and attitudes on gender inequity, validated in Tanzania and Ghana, with good reliability in African settings. Domains include violence, sexual relationships, reproductive health and disease prevention, and domestic chores and daily life items. Higher scores indicate more inequitable gender attitudes. Possible score range = 1-3.

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere School of Public Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
All collected quantitative IPD. For the qualitative data, we will limit the sharing to include the sharing of codes, themes, and interview guides. We will not share transcripts or segments of coded transcripts, given difficulty to fully de-identify qualitative data, to protect participant privacy and confidentiality.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be will shared at the time of publication or at the end of data analysis (anticipated by May 15, 2029)
Access Criteria: Data, data analysis code, and associated meta-data (data collection tools that generated the data) will be made accessible in the NICHD Data and Specimen Hub (DASH), a centralized resource that allows researchers to share and access de-identified data from studies funded by NICHD.

REFERENCES:
- [Background] Sileo KM, Muhumuza C, Wanyenze RK, Kershaw TS, Sekamatte S, Lule H, Kiene SM. A pilot quasi-experimental controlled trial of a community-based, multilevel family planning intervention for couples in rural Uganda: evidence of feasibility, acceptability, and effect on contraceptive uptake among those with an unmet need for family planning. Contraception. 2023 Sep;125:110096. doi: 10.1016/j.contraception.2023.110096. Epub 2023 Jun 22. PMID 37355086